CLINICAL TRIAL: NCT04140227
Title: A Phase 3, Multi-Center, Open-Label, Single-Arm Extension Clinical Trial to Assess the Extended Long-Term Safety and Tolerability of NOV03 (Perfluorohexyloctane) in Subjects Who Completed Trial NVU-003 (Kalahari Study)
Brief Title: Long-Term Safety and Tolerability of NOV03 (Perfluorohexyloctane) in Subjects Who Completed Trial NVU-003 (Kalahari Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVU-004 (Kalahari)
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Results first posted 2023-12-29 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2022-01

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NOV03 4 times daily (QID) (Experimental): 100% Perfluorohexyloctance solution 4 times daily (QID)
  Interventions: Drug: NOV03

INTERVENTIONS:
Drug: NOV03 — 100% Perfluorohexyloctane

SUMMARY:
The objectives of this trial are to evaluate the safety and tolerability of perfluorohexyloctane (NOV03) ophthalmic solution during long-term use in subjects with Dry Eye Disease (DED) associated with MGD (Meibomian Gland Dysfunction).

Further objective is to evaluate the efficacy of perfluorohexyloctane (NOV03) solution during long-term use in subjects with DED associated with MGD.

DETAILED DESCRIPTION:
The objectives of this trial are to evaluate the safety and tolerability of perfluorohexyloctane (NOV03) ophthalmic solution during long-term use in subjects with Dry Eye Disease (DED) associated with MGD (Meibomian Gland Dysfunction).

Further objective is to evaluate the efficacy of perfluorohexyloctane (NOV03) solution during long-term use in subjects with DED associated with MGD.

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF (Informed Consent Form)
* Subject-reported history of Drye Eye Disease (DED) in both eyes
* Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

* Women who are pregnant, nursing or planning pregnancy
* Unwillingness to submit a blood pregnancy test at screening and the last visit (or early termination visit) if of childbearing potential, or unwillingness to use acceptable means of birth control
* Clinically significant slit-lamp findings or abnormal lid anatomy at screening
* Ocular/peri-ocular malignancy
* History of herpetic keratitis
* Active ocular allergies or ocular allergies that are expected to be active during the study
* Ongoing ocular or systemic infection
* Wear contact lenses within 1 month prior to screening or anticipated use of contact lenses during the study
* Intra-ocular surgery or ocular laser surgery within the previous 6 months, or have planned ocular and/or lid surgeries over the study period
* Presence of uncontrolled systemic diseases
* Presence of known allergy and/or sensitivity to the study drug or saline components
* Use of any topical steroids treatments, topical cyclosporine, lifitegrast, serum tears or topical anti-glaucoma medication within 2 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2022-01-05 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Bausch Health
Locations (28):
- United States (28):
  - Bausch Site 124, Birmingham, Alabama
  - Bausch Site 125, Scottsdale, Arizona
  - Bausch Site 110, Glendale, California
  - Bausch Site 121, Long Beach, California
  - Bausch Site 102, Mission Hills, California
  - Bausch Site 101, Newport Beach, California
  - Bausch Site 116, Rancho Cordova, California
  - Bausch Site 103, Torrance, California
  - Bausch Site 123, Torrance, California
  - Bausch Site 127, Danbury, Connecticut
  - Bausch Site 129, Fort Myers, Florida
  - Bausch Site 115, Jacksonville, Florida
  - Bausch Site 106, Largo, Florida
  - Bausch Site 117, Tampa, Florida
  - Bausch Site 108, Lake Villa, Illinois
  - Bausch Site 112, Indianapolis, Indiana
  - Bausch Site 119, Edgewood, Kentucky
  - Bausch Site 126, Winchester, Massachusetts
  - Bausch Site 113, Kansas City, Missouri
  - Bausch Site 111, St Louis, Missouri
  - Bausch Site 128, Slingerlands, New York
  - Bausch Site 114, Raleigh, North Carolina
  - Bausch Site 122, Cranberry Township, Pennsylvania
  - Bausch Site 107, Memphis, Tennessee
  - Bausch Site 109, Nashville, Tennessee
  - Bausch Site 120, El Paso, Texas
  - Bausch Site 104, Lakeway, Texas
  - Bausch Site 118, San Antonio, Texas

REFERENCES:
- [Derived] Protzko EE, Segal BA, Korenfeld MS, Krosser S, Vittitow JL. Long-Term Safety and Efficacy of Perfluorohexyloctane Ophthalmic Solution for the Treatment of Patients With Dry Eye Disease: The KALAHARI Study. Cornea. 2024 Sep 1;43(9):1100-1107. doi: 10.1097/ICO.0000000000003418. Epub 2023 Nov 3. PMID 37921522

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NOV03 4 Times Daily (QID)
Started | 256
Completed | 208
Not Completed | 48
Not completed — Withdrawal by Subject | 26
Not completed — Lost to Follow-up | 8
Not completed — Adverse Event | 8
Not completed — Death | 1
Not completed — Other | 3
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Groups:
- Single-arm Open Label: single-arm open label
Arm/Group | Single-arm Open Label
Number analyzed (Participants) | 208
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (13.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 43
  White | 133
  More than one race | 0
  Unknown or Not Reported | 1
Type of Eyes [Count of Participants; unit: Participants]
  Right Eye | 121
  Left Eye | 87

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ocular and Non-ocular Adverse Events
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | NOV03 4 Times Daily (QID)
Number analyzed (Participants) | 208
Participants
  At Least 1 TEAE Ocular and non-Ocular | 69
  At Least 1 IP-related TEAE Ocular and non-Ocular | 14
  At Least 1 SAE Ocular and non-Ocular | 1
  TEAE that led to Drug Withdrawal | 9

ADVERSE EVENTS:
Time Frame: AE information was captured during the duration of the study of 1 year
Arm/Group | NOV03 4 Times Daily (QID)
All-Cause Mortality (participants affected / at risk) | 1/208
Serious Adverse Events (participants affected / at risk) | 10/208
Other Adverse Events (participants affected / at risk) | 44/208
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOV03 4 Times Daily (QID) (N=208)
Severe Gastric Cancer (Gastrointestinal disorders) | 1 (1)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypoglcaemia (Metabolism and nutrition disorders) | 1 (1)
femur fracture (Injury, poisoning and procedural complications) | 1 (1)
radius fracture (Injury, poisoning and procedural complications) | 1 (1)
tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
ulna fracture (Injury, poisoning and procedural complications) | 1 (1)
transient ischaemic attack (Cardiac disorders) | 1 (1)
schizophrenia (Psychiatric disorders) | 1 (1)
spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cerebrovascular accident (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NOV03 4 Times Daily (QID) (N=208)
Sinusitis (Infections and infestations) | 2
COVID-19 (Infections and infestations) | 6
Urinary Tract Infection (Infections and infestations) | 2
Hypertension (Vascular disorders) | 4
Vitreous detachment (Eye disorders) | 4
Conjuctivitis allergic (Eye disorders) | 3
Lacrimation increased (Eye disorders) | 3
Vision blurred (Eye disorders) | 3
Dry eye (Eye disorders) | 2
Instillation site pain (General disorders) | 2
Hordeolum (Infections and infestations) | 2
Chalazion (Eye disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Neuralgia (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT04140227/Prot_SAP_000.pdf